CLINICAL TRIAL: NCT02135744
Title: Pre-Discharge Bundle for Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease to Reduce Readmissions and Emergency Department Visits: a Randomized, Controlled Trial.
Brief Title: Pre-Discharge Bundle for Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease to Reduce Readmissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jeffrey Jennings, Staff Physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6174
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Readmissions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Group of patients undergo standard care as determined by the primary inpatient team
- Bundle (Experimental): Group of patients that receive the screening and educational tool
  Interventions: Behavioral: Bundle tool

INTERVENTIONS:
Behavioral: Bundle tool — Tool consists of 1. screening measures to identify the presence of various risk factors for COPD exacerbations and 2. Educational components for the disease of COPD.
  Arms: Bundle

SUMMARY:
Hospital readmissions for acute exacerbations of chronic obstructive pulmonary disease (AECOPD) pose burdens to the healthcare system and patients. The aim of this study was to determine whether a screening and educational tool, administered prior to discharge, would result in a decrease in the rate of hospital readmissions.

DETAILED DESCRIPTION:
Hospital readmissions for acute exacerbations of chronic obstructive pulmonary disease (AECOPD) pose burdens to the healthcare system and patients. A current gap in knowledge is whether a pre-discharge screening and educational tool, administered to patients with COPD, reduces readmissions and emergency department (ED) visits.

A single center, randomized trial of patients admitted with AECOPD. Patients will be randomized to control (standard care) or "bundle" group in which patients receive smoking cessation counseling, screening for gastroesophageal reflux disease and depression or anxiety, standardized inhaler teaching, and a 48-hour post-discharge phone call.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD with the presence of an AECOPD
* Age > 40
* Current or ex-smoker with history of at least 20 pack-years

Exclusion Criteria:

* Past history of asthma, interstitial lung disease, bronchiectasis, presence of airway hardware (e.g. tracheal stents or tracheotomy), lung cancer, any other cancer with a life expectancy of less than 1 year
* Presence of a language barrier
* Residence in a nursing home
* Intensive care unit stay during the current admission
* Delirium or dementia.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
30 day readmission rate | 30 days
  Time until readmission or ER visit, 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Jennings JH, Thavarajah K, Mendez MP, Eichenhorn M, Kvale P, Yessayan L. Predischarge bundle for patients with acute exacerbations of COPD to reduce readmissions and ED visits: a randomized controlled trial. Chest. 2015 May;147(5):1227-1234. doi: 10.1378/chest.14-1123. PMID 25940250